CLINICAL TRIAL: NCT05478850
Title: An Observational Cohort Study of Inadvertent Hypothermia or Hyperthermia in Pediatric Radiotherapy Practices Under Anesthesia
Brief Title: Inadvertent Hypothermia or Hyperthermia in Pediatric Radiotherapy Practices Under Anesthesia
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Betül Güven, Principle Investigator, Ankara City Hospital Bilkent
Other Study IDs: E1-22-2700
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-07

CONDITIONS: Hypothermia; Anesthesia; Hyperthermia, Anesthesia Related; Radiotherapy Side Effect; Childhood Cancer
Keywords: Hypothermia; Anesthesia; Hyperthermia, Anesthesia Related; Radiotherapy Side Effect; Childhood Cancer
MeSH Terms: conditions — Hypothermia; Malignant Hyperthermia; Radiation Injuries; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiotherapy under anesthesia
  Interventions: Procedure: radiotherapy under anesthesia

INTERVENTIONS:
Procedure: radiotherapy under anesthesia — Body temperature change will be investigated before the procedure and during recovery in Radiotherapy patients who need anesthesia due to childhood malignancies.

SUMMARY:
In prospective, observational cohort study, changes in body temperature will be investigated before the procedure and during recovery in Radiotherapy patients aged 0-18 years who need sedation due to childhood malignancies.

The aims of this study were to measure the incidence and magnitude of changes in body temperature in children undergoing sedation or general anesthesia for Radiotherapy, and to determine their effects on the recovery process.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing radiotherapy under anesthesia

Exclusion Criteria:

* family refusal to participate,
* chronic nausea and vomiting complaints,
* active infection,
* apnea history,
* cardiac disease, kidney and liver failure,
* anomalies that may cause difficult airway,
* metabolic diseases,
* neurological or muscular diseases.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients undergoing radiotherapy under anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
body temperature change among 2 time period | time from before radiotherapy to the end of radiotherapy
  non-contact body temperature measured on forehead
recovery time from anesthesia | the time from end of radiotherapy to discharging
  Time from the end of the procedure until the Modified Steward score ≥ 8 in the patient recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Betül Güven Aytaç, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided